CLINICAL TRIAL: NCT00370539
Title: Combined PDT and Intravitreal Bevacizumab vs Combination of PDT, Intravitreal Bevacizumab and Triamcinolone for Neovascular AMD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8542
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-11

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Photodynamic therapy,; Bevacizumab,; Triamcinolone,; Age-related macular degeneration,; Choroidal neovascular membrane
MeSH Terms: conditions — Macular Degeneration | interventions — Verteporfin; Bevacizumab; Triamcinolone Acetonide

INTERVENTIONS:
Drug: verteporfin, bevacizumab, triamcinolone acetonide

SUMMARY:
To compare the efficacy and safety of photodynamic therapy (PDT) combined with intravitreal bevacizumab versus combination of photodynamic therapy , intravitreal bevacizumab and intravitreal triamcinolone for neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

* Cases of active neovascular AMD with visual acuity of 20/400- 20/40

Exclusion Criteria:

* History of glaucoma or ocular hypertension
* Disciform scar

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-09; Study Completion 2006-11

PRIMARY OUTCOMES:
Visual acuity

SECONDARY OUTCOMES:
Central macular thickness
Leakage in fluorescein angiography
Intraocular pressure
Anterior chamber reaction

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh, MD, Tehran, Tehran Province, Iran